CLINICAL TRIAL: NCT01242163
Title: Application of Chemical Sensors for Diagnosis of Inflammatory Bowel Diseases and Irritable Bowel Syndrome by Respiratory Samples
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Dr Amir Karban, Rambam Medical Center
Other Study IDs: 0481-10CTIL
Record Dates: First submitted 2010-11-14; First posted 2010-11-16 (Estimated); Last update posted 2010-11-23 (Estimated); Status verified 2010-10

CONDITIONS: Inflammatory Bowel Diseases; Irritable Bowel Syndrome
MeSH Terms: conditions — Inflammatory Bowel Diseases; Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Experiated lung air
Oversight: Data Monitoring Committee: No

SUMMARY:
Discriminating irritable bowel syndrome (IBS) from inflammatory bowel disease (IBD), especially with mild disease activity, is common clinical challenge. Most of the patients with suspected IBS have to go invasive procedures (colonoscopy/gastroscopy). In order to avoid invasive investigations, there is a search for noninvasive markers with the capacity to distinguish between IBS and IBD. Dr Hossam Haick (Department of Chemical Engineering, Technion) developed a system that combines nano-metals produced in his laboratory with electrical devices (transistors). The combination between a nanomaterial and an electrical transistor induces a change in its electrical behavior upon exposure to the material being examined; that is, a change in its electrical properties. The change in its electrical behavior is translated into a computerized graphic signal.

The electronic nose is composed of an air pump, a filter for filtering external contaminants and an array of sensors. Each sensor transmits a signal according to the materials it "knows" how to identify. Thus, it is possible to characterize most of the substance families characteristic of a certain disease, and the same system is designed for differential diagnosis of different diseases.

The purpose of the investigators study is to use the "electronic nose" to find bio-markers that will help to diagnose IBD and IBS without using invasive procedures.

The plan is to collect 200 samples (50 IBS' 50 Crohn's disease, 50 ulcerative colitis and 50 controls). The patients included in the study will undergo an evaluation by a gastroenterologist after signing an informed consent and will answer a questionnaire.

The samples will analyzed in the laboratory of Dr. Haick.

DETAILED DESCRIPTION:
The plan is to collect 200 samples (50 IBS' 50 Crohn's disease, 50 ulcerative colitis and 50 controls). The patients included in the study will undergo an evaluation by a gastroenterologist after signing an informed consent and will answer a questionnaire.

The samples will analyzed in the laboratory of Dr. Haick.

ELIGIBILITY:
Inclusion Criteria:

* Patinets with IBD or IBS

Exclusion Criteria:

* Age under 18 y/o pregnancy, malignant and infectious diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Inflammtory bowel Diseases and IBS
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2010-12; Study Completion 2012-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Amir Karban, MD, Principal Investigator — Rambam Medical Center, Haifa, Israel